CLINICAL TRIAL: NCT04046497
Title: Early-phase Schizophrenia: Practice-based Research to Improve Outcomes (ESPRITO) - Using Artificial Intelligence to Measure Adherence to Oral Medication
Brief Title: Artificial Intelligence to Measure Adherence to Oral Medication
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-0307-ZHH
Record Dates: First submitted 2019-07-01; First posted 2019-08-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: First Episode Psychosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone App (Experimental): artificial intelligence (AI) smartphone app to provide support for medication adherence
  Interventions: Other: Smartphone App
- Usual Care (Active Comparator): Usual care provided at CSC clinic
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Smartphone App — artificial intelligence (AI) smartphone app to provide support for medication adherence
  Arms: Smartphone App
Other: Usual Care — Usual Care provided by CSC clinic
  Arms: Usual Care

SUMMARY:
The aims of this project is to use an artificial intelligence (AI) smartphone app to provide support for medication adherence by patients with first episode psychosis.

DETAILED DESCRIPTION:
The challenge of oral medication adherence in first-episode psychosis (as in any potentially chronic illness) is enormous, and numerous studies have linked non-adherence to increased rates of relapse/ hospitalization. Determining whether a patient is adhering to medication is a challenge. Pill counts, pharmacy records, technology-assisted monitoring, biological assays, and a range of self-report and interviewer-rated scales have been employed. In other areas of medicine such as antiretroviral treatment Direct Observation of Treatment (DOT) has been employed with excellent success both in monitoring and demonstrated improvement of important clinical outcomes. DOT is clearly not feasible in community settings. An artificial Intelligence (AI) platform that can be downloaded as an application onto a smart phone app represents a novel approach to offering DOT to support participant oral medication adherence and thereby improve outcomes. Aims of the project are: 1) to document acceptability to patients of the AI smartphone app based upon participation in the study and 2) to compare rates of hospitalization and emergency room visits between participants who receive the AI smartphone app with participants who receive standard care.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a CSC program
* Prescribed an oral antipsychotic

Exclusion Criteria:

* none

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Service Utilization Report Form | 12 months
  Provides participant utilization of psychiatric ER visits or psychiatric hospitalization

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Citrus Health, Hialeah, Florida
  - InterAct, Grand Rapids, Michigan
  - InterAct of Michigan, Kalamazoo, Michigan
  - Red Rock, Oklahoma City, Oklahoma
  - Family and Children's Services, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No